CLINICAL TRIAL: NCT02800759
Title: The Minimal Effective Dose of Cis-9-cetylmyristoleate (CMO) in Persons Presenting With Knee Joint Pain
Brief Title: Effect of Cis-9-cetylmyristoleate in Sub-healthy Subjects Presenting With Knee Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Clinical Associate Professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1307-098-506
Record Dates: First submitted 2016-06-08; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Knee Pain Intermittent
MeSH Terms: interventions — cetyl myristoleate; Reppal PES 100

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 100% of JOINTRUS® (Active Comparator): After randomization, 100% dose of JOINTRUS® is taken per day for 3 months in 7 sub-healthy persons >18 years of age and knee joint pain with a 0-10 numerical rating scale (NRS) pain score ≤ 4. This study included a 7-day baseline screening period (Visit 1) and was followed by randomization (Visit 2), a 12-week ingestion period with clinic visits at week 4 (Visit 3), 8 (Visit 4), and 12 (Visit 5) after starting ingestion, and a 4-week post-ingestion safety follow-up. The pain intensity, functional disability state and change in the general status were assessed for a 12-week ingestion period.
  Interventions: Dietary Supplement: JOINTRUS®
- 80% of JOINTRUS® (Active Comparator): After randomization, 80% dose of JOINTRUS® was taken per day for 3 months in 7 sub-healthy persons >18 years of age and knee joint pain with a 0-10 numerical rating scale (NRS) pain score ≤ 4. This study included a 7-day baseline screening period (Visit 1) and was followed by randomization (Visit 2), a 12-week ingestion period with clinic visits at week 4 (Visit 3), 8 (Visit 4), and 12 (Visit 5) after starting ingestion, and a 4-week post-ingestion safety follow-up. The pain intensity, functional disability state and change in the general status were assessed for a 12-week ingestion period.
  Interventions: Dietary Supplement: 80% dose of JOINTRUS®
- 62.4% of JOINTRUS® (Active Comparator): After randomization, 62.4% dose of JOINTRUS® was taken per day for 3 months in 7 sub-healthy persons >18 years of age and knee joint pain with a 0-10 numerical rating scale (NRS) pain score ≤ 4. This study included a 7-day baseline screening period (Visit 1) and was followed by randomization (Visit 2), a 12-week ingestion period with clinic visits at week 4 (Visit 3), 8 (Visit 4), and 12 (Visit 5) after starting ingestion, and a 4-week post-ingestion safety follow-up. The pain intensity, functional disability state and change in the general status were assessed for a 12-week ingestion period.
  Interventions: Dietary Supplement: 62.4% dose of JOINTRUS®
- Starch 100% (Placebo Comparator): After randomization, starch 100% was taken per day for 3 months in 7 sub-healthy persons >18 years of age and knee joint pain with a 0-10 numerical rating scale (NRS) pain score ≤ 4. This study included a 7-day baseline screening period (Visit 1) and was followed by randomization (Visit 2), a 12-week ingestion period with clinic visits at week 4 (Visit 3), 8 (Visit 4), and 12 (Visit 5) after starting ingestion, and a 4-week post-ingestion safety follow-up. The pain intensity, functional disability state and change in the general status were assessed for a 12-week ingestion period.
  Interventions: Dietary Supplement: Starch 100%

INTERVENTIONS:
Dietary Supplement: JOINTRUS® — 100% Fatty acid compound with 12.5% Cis-9-cetylmyristoleate
  Other Names: 100% Fatty acid compound with 12.5% Cis-9-cetylmyristoleate
  Arms: 100% of JOINTRUS®
Dietary Supplement: 80% dose of JOINTRUS® — 80% Fatty acid compound with 12.5% Cis-9-cetylmyristoleate
  Other Names: 80% Fatty acid compound with 12.5% Cis-9-cetylmyristoleate
  Arms: 80% of JOINTRUS®
Dietary Supplement: 62.4% dose of JOINTRUS® — 62.4% Fatty acid compound with 12.5% Cis-9-cetylmyristoleate
  Arms: 62.4% of JOINTRUS®
Dietary Supplement: Starch 100% — 0% Fatty acid compound with 12.5% Cis-9-cetylmyristoleate
  Arms: Starch 100%

SUMMARY:
Cis-9-cetylmyristoleate (CMO) is a naturally occurring fatty acid complex (FAC). Nutraceuticals containing CMO are used to improve knee pain despite the lack of placebo-controlled studies in humans. The aim of the double-blind controlled clinical trial is to explore the minimal effective dose of CMO for relieving knee joint pain.

DETAILED DESCRIPTION:
Methods: Twenty-eight subjects, who are clinically or radiologically diagnosed as having mild degree arthritic knee joint pain, are randomized into 3 groups; Groups A, B, C that contained 100%, 80%, and 62.4% of fatty acid component with 12.5% of Cis-9-cetylmyristoleate (CMO), and control Group D (starch 100%). The pain intensity, functional disability state and change in the general status were assessed for a 12-week ingestion period.

ELIGIBILITY:
Inclusion Criteria:

* sub-healthy persons >18 years of age and knee joint pain with a 0-10 numerical rating scale (NRS) pain score ≤ 4.

Exclusion Criteria:

* current medication use related to arthritis;
* current use of FAC containing products;
* clinical or radiological diagnosis as moderate degree arthritis accompanied by peri-articular spur formation, irregular joint margin, and/or subchondral cyst;
* previous history of knee surgery;
* pregnant, breastfeeding, or practicing contraception with reliable methods, or not accepting our guidelines during the research periods;
* major pain other than knee joint pain;
* current treatment of gastritis or gastric ulcer;
* abnormal screening laboratory results;
* major cardiac, renal disease, or disability that could affect adverse effect assessment or interfere with study completion when enrolled;
* history of major procedures or operations that might affect study results;
* enrollment in another clinical trial or human application testing; and
* judged as unsuitable for human application testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
CHANGE of Pain | change from baseline at 3 months
  using the NRS score, composed of an 11-point scale from 0 (no pain) to 10 (the worst pain possible)

SECONDARY OUTCOMES:
difference in NRS pain score from baseline within groups | at 1-month follow-up, at 2-month follow-up, and at 3-month follow-up
change of the WOMAC score | change from baseline at 3 months
  using the Korean version of WOMAC
Global Impression of Change | at 3-month follow-up
  a scale ranging from 1 (very much improved) to 7 (very much worse).

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Thiem U, Lamsfuss R, Gunther S, Schumacher J, Baker C, Endres HG, Zacher J, Burmester GR, Pientka L. Prevalence of self-reported pain, joint complaints and knee or hip complaints in adults aged >/= 40 years: a cross-sectional survey in Herne, Germany. PLoS One. 2013 Apr 30;8(4):e60753. doi: 10.1371/journal.pone.0060753. Print 2013. PMID 23646102
- [Background] Nguyen US, Zhang Y, Zhu Y, Niu J, Zhang B, Felson DT. Increasing prevalence of knee pain and symptomatic knee osteoarthritis: survey and cohort data. Ann Intern Med. 2011 Dec 6;155(11):725-32. doi: 10.7326/0003-4819-155-11-201112060-00004. PMID 22147711
- [Background] Pereira D, Peleteiro B, Araujo J, Branco J, Santos RA, Ramos E. The effect of osteoarthritis definition on prevalence and incidence estimates: a systematic review. Osteoarthritis Cartilage. 2011 Nov;19(11):1270-85. doi: 10.1016/j.joca.2011.08.009. Epub 2011 Aug 24. PMID 21907813
- [Background] Zhang W, Doherty M, Arden N, Bannwarth B, Bijlsma J, Gunther KP, Hauselmann HJ, Herrero-Beaumont G, Jordan K, Kaklamanis P, Leeb B, Lequesne M, Lohmander S, Mazieres B, Martin-Mola E, Pavelka K, Pendleton A, Punzi L, Swoboda B, Varatojo R, Verbruggen G, Zimmermann-Gorska I, Dougados M; EULAR Standing Committee for International Clinical Studies Including Therapeutics (ESCISIT). EULAR evidence based recommendations for the management of hip osteoarthritis: report of a task force of the EULAR Standing Committee for International Clinical Studies Including Therapeutics (ESCISIT). Ann Rheum Dis. 2005 May;64(5):669-81. doi: 10.1136/ard.2004.028886. Epub 2004 Oct 7. PMID 15471891
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, part I: critical appraisal of existing treatment guidelines and systematic review of current research evidence. Osteoarthritis Cartilage. 2007 Sep;15(9):981-1000. doi: 10.1016/j.joca.2007.06.014. Epub 2007 Aug 27. PMID 17719803
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage. 2008 Feb;16(2):137-62. doi: 10.1016/j.joca.2007.12.013. PMID 18279766
- [Background] Zhang W, Nuki G, Moskowitz RW, Abramson S, Altman RD, Arden NK, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis: part III: Changes in evidence following systematic cumulative update of research published through January 2009. Osteoarthritis Cartilage. 2010 Apr;18(4):476-99. doi: 10.1016/j.joca.2010.01.013. Epub 2010 Feb 11. PMID 20170770
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672